CLINICAL TRIAL: NCT02602951
Title: 4D FLOW: Feasibility Study of a Sequence 4D of Flow Applied to the Cervico-encephalic Vascular Pathologies
Acronym: 4D-FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D15-P006
Record Dates: First submitted 2015-10-06; First posted 2015-11-11 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Cerebro-vascular Disease
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Pilot subjects
  Interventions: Other: Pilot MRI program
- Patients (Experimental): Patients with an intracranial disorder or needing a supraaortic trunk MRA
  Interventions: Other: MRI with 4D Flow sequence

INTERVENTIONS:
Other: Pilot MRI program — Pilot MRI program
  Arms: Control
Other: MRI with 4D Flow sequence — MRI with 4D Flow sequence
  Arms: Patients

SUMMARY:
The dynamic angio-MR sequences with injection of contrast (CE ARM) allow the study of the vascular anatomy. These sequences, widely used in clinical routine have shown their utility, in particular in the detection of the cerebrovascular diseases. The 4D flow MR sequences allow to quantify arterial parameters such as the speed of the circulating flow. By allowing an anatomical analysis and a functional analysis of quantitative parameters, 4D flow MR sequences could replace 1/ the currently used dynamic MRA sequences that are less precise in term of spatial and temporal resolution; 2/ the invasive exploration by DSA for the detection of vascular lesion and complete the exploration of the cervico-encephalic vascular pathologies by providing hemodynamical measures not yet accessible in clinical settings.

In this context, the aim of the study is to evaluate the feasibility and the clinical usefulness of this 4D Flow technique to image brain vascular disorders including steno occlusive disorders. The evaluation will include several steps: 1/ optimization of acquisition parameters for the cranio-cervical arteries; 2/ comparison of two strategies for the post-processing 3/ feasibility for imaging of brain vascular disorders.

DETAILED DESCRIPTION:
The dynamic angio-MR sequences with injection of contrast (CE ARM) allow the study of the vascular anatomy. These sequences, widely used in clinical routine have shown their utility, in particular in the detection of the cerebrovascular diseases. The 4D flow MR sequences allow to quantify arterial parameters such as the speed of the circulating flow. By allowing an anatomical analysis and a functional analysis of quantitative parameters, 4D flow MR sequences could replace 1/ the currently used dynamic MRA sequences that are less precise in term of spatial and temporal resolution; 2/ the invasive exploration by DSA for the detection of vascular lesion and complete the exploration of the cervico-encephalic vascular pathologies (arterio-venous deformations, cervical or intra-cranial stenoses, intra-cranial aneurysms) by providing hemodynamical measures not yet accessible in clinical settings.

In this context, the aim of the study is to evaluate the feasibility and the clinical usefulness of this 4D Flow technique to image brain vascular disorders including steno occlusive disorders. The evaluation will include several steps: 1/ optimization of acquisition parameters for the cranio-cervical arteries; 2/ comparison of two strategies for the post-processing 3/ feasibility for imaging of brain vascular disorders.

STUDY HYPOTHESIS & AIMS The investilgators hypothesized that, once optimized for brain and cervical acquisition, 4D flow MRA will provides quantitative information not available with other routinely available dynamic MR sequences. The main goal of this study is to demonstrate the feasibility of a non-invasive evaluation of hemodynamics (quantitative speed measurements and flow tracking) in neuro applications using the 4D Flow prototype. The secondary goal is to compare parameters derived from 4D Flow prototype using two post-processing pipelines.

4D Flow images will be compared to other available hemodynamic information obtained as part of the routine clinical care in order to assess whether additional clinically relevant information can be extracted.

The study of the arterio-venous deformations and the study of the supraaortic trunks require the realization of MRI sequences with injection of Gd during a clinical protocol of routine. The sequence added at the end of protocol does not modify the injection with clinical purpose.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patient of 18 years old and more
* Patient reffered to the imaging department for a MRI for the exploration of a cervical or intracranial vascular disease (cervical stenosis, arterio-venous malformation)
* Patient whose MRI requires an injection of gadolinium
* Patient with insurance
* Informed consent

Experimental subjects:

* Absence of known cerebral or arterial pathology. Absence of MR contraindication
* 18 years old or more

Exclusion Criteria:

* Emergency situation: patient in an urgent situation care
* Contraindications to the administration of Gadolinium (patients only)
* Contraindications to MRI :

cardiac or neuronal stimulating device, ferromagnetic surgical Clips, cochlear Implants, metallic intraocular Foreign bodies or in the nervous system

* Claustrophobia
* Pregnant Women
* Subjects deprived of freedom by court order or administration staff
* Major Subjects protected by the law
* Known Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting linear flow conditions assessed by the visual analysis of computed streamlines visualisation | through study completion, an average of 12 months
  Flow tracking (clinical utility on the basis of qualitative criteria).

SECONDARY OUTCOMES:
Speed measurement (m/s) of velocitymeasured in the crossection of vessels. | through study completion, an average of 12 months
  Measures of speeds
Flow aliasing within the vessels. | through study completion, an average of 12 months
  criteria for image Quality (Image quality will be centered on the presence or absence of flow aliasing within the vessels.)

CONTACTS AND LOCATIONS:
Overall Officials: Myriam EDJLALI, MD, Study Director — Centre Hospitalier Sainte-Anne
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France